CLINICAL TRIAL: NCT04274894
Title: 24-Hour Ambulatory Blood Pressure Monitoring Study in Hypogonadal Men Receiving Testosterone Replacement Therapy
Brief Title: A Study of the Effect of Topical Testosterone Replacement Therapy on Blood Pressure in Adult Male Participants With Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19-161
Record Dates: First submitted 2020-02-17; First posted 2020-02-18 (Actual); Results first posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-11

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Testosterone Replacement Therapy; AndroGel
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AndroGel 1.62% (Experimental): AndroGel 1.62% was applied topically once daily in the morning beginning at the Day 1 Visit after confirmed valid ambulatory blood pressure monitoring (ABPM) assessment and was applied at approximately the same time each day after that during the study, for approximately 16 weeks. The starting dose of AndroGel 1.62% was 40.5 mg of T (2 pump actuations, applied to the upper arms and shoulders) and was titrated up or down by 20.25 mg or remained the same as assessed by morning serum T levels at Weeks 2 and 4.
  Interventions: Drug: AndroGel 1.62%

INTERVENTIONS:
Drug: AndroGel 1.62% — AndroGel 1.62% was packaged in pump bottles with quantities sufficient to accommodate study design and could have been dose adjusted between a minimum of 20.25 mg of T (1 pump actuation) and a maximum of 81.0 mg of testosterone (4 pump actuations). For the first study drug administration at the Day 1 Visit, and also at Week 2, Week 4, Week 16 ambulatory blood pressure monitoring (ABPM,) and End of Treatment Visits, participants applied the study drug while on site so that the site staff could observe the proper administration of study drug. If participants forgot to apply their AndroGel 1.62% dose at their regularly scheduled dosing time, they were to take the next dose at the next dosing time.
  Other Names: Testosterone gel

SUMMARY:
Hypogonadism is an endocrine disorder characterized by absent or deficient testosterone levels along with signs and symptoms of androgen deficiency, including delayed development or regression of sexual characteristics, impaired sexual function and sense of well-being, depressed mood, decreased muscle strength associated with loss of muscle mass and reduced bone mineral density. AndroGel 1.62% has demonstrated its ability to increase total testosterone levels in the blood by absorption of testosterone through the skin when applied topically. This study evaluated the effect of AndroGel 1.62% on systolic blood pressure using ambulatory blood pressure monitoring in hypogonadal men who used testosterone replacement therapy.

AndroGel 1.62% is a drug used for the treatment of hypogonadism, which is associated with low or no testosterone. This was an open-label study which means that both the study doctor and study participants knew what drug and what dose is being used. All participants in this study were in the same group, called a treatment arm. Adult male participants with hypogonadism were enrolled and received AndroGel 1.62%. This was a multi-center study with 190 participants enrolled (initially planned) in approximately 45 sites in the United States to yield 171 subjects in the per protocol (PP) population. A blinded sample size re-estimation (BSSR) was performed when around 70% of the planned subjects in the PP population had completed the end of treatment visit. Sample size was increased at BSSR and 246 participants were actually enrolled.

Participants received daily topical gel doses of AndroGel 1.62% for approximately 16 weeks.

There may have been a higher burden for participants in this study compared to standard of care. Participants attended 8 study visits during the course of the study at a hospital or clinic and received 2 study phone calls. The effect of the treatment was checked by medical assessments, blood tests (including pharmacokinetic sampling), and 24-hour blood pressure monitors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypogonadism with the presence of at least one of the following symptoms that may be related to low testosterone values and is/are consistent with hypogonadism:

  * Decreased sexual desire or libido
  * Decreased spontaneous erections (e.g. morning erections)
  * Decreased energy or fatigue/feeling tired
  * Low mood or depressed mood
  * Loss of body (axillary and pubic) hair or reduced shaving
  * Hot flashes AND
* Confirmed by 2 serum testosterone levels < 300 ng/dL by blood samples drawn at least 48 hours apart. These samples should be obtained between 5 am and 11 am local time.
* Blood pressure >100/60 mmHg and <140/90 mmHg

Exclusion Criteria:

* Unprovoked deep vein thrombosis (DVT), unprovoked pulmonary embolism (PE), or known thrombophilia
* Polycythemia vera or secondary polycythemia, such as polycythemia due to untreated sleep apnea or severe chronic obstructive pulmonary disease
* Prostate or breast cancer
* Any active malignancy
* Clinically significant medical conditions or any other reason that the investigator determines would interfere with participation in this study or would make the participant an unsuitable candidate to receive study drug
* Work night shifts or is otherwise required to perform strenuous manual labor while wearing the Ambulatory Blood Pressure Monitor (ABPM).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (45):
- United States (45):
  - G & L Research, LLC /ID# 216793, Foley, Alabama
  - NewportNativeMD, Inc. /ID# 216992, Newport Beach, California
  - Valley Renal Medical Group Research /ID# 216321, Northridge, California
  - West Coast Research LLC /ID# 216813, San Ramon, California
  - Lynn Institute of Denver /ID# 216863, Aurora, Colorado
  - Innovative Research of West Florida /ID# 216364, Clearwater, Florida
  - Seidman Clinical Trials,Delray /ID# 216794, Delray Beach, Florida
  - Invesclinic, U.S., LLC /ID# 216778, Fort Lauderdale, Florida
  - Indago Research and Health Cen /ID# 216319, Hialeah, Florida
  - Care Partners Clinical Research /ID# 216773, Jacksonville, Florida
  - Pharmax Research Clinic /ID# 216343, Miami, Florida
  - Care Research center Inc. /ID# 216367, Miami, Florida
  - West Orange Endocrinology /ID# 217106, Ocoee, Florida
  - North Georgia Clinical Research /ID# 216864, Woodstock, Georgia
  - Solaris Clinical Research /ID# 216772, Meridian, Idaho
  - Loretto Hospital.Affnity Clinical Research Institute /ID# 216884, Chicago, Illinois
  - Affinity Clinical Research /ID# 216807, Oak Brook, Illinois
  - Investigative Clinical Research of Indiana, LLC /ID# 216943, Elwood, Indiana
  - Iowa Diabetes and Endocrinology Research Center /ID# 216316, West Des Moines, Iowa
  - PRN Professional Research Network of Kansas, LLC /ID# 216805, Wichita, Kansas
  - The Research Grp of Lexington /ID# 216451, Lexington, Kentucky
  - Centennial Medical Group /ID# 216340, Elkridge, Maryland
  - Advanced Biomedical Research of America /ID# 216797, Las Vegas, Nevada
  - Amici Clinical Research /ID# 216779, Warren Township, New Jersey
  - NM Clinical Research & Osteoporosis Center, Inc /ID# 216808, Albuquerque, New Mexico
  - AccuMed Research Associates /ID# 216775, Garden City, New York
  - Randolph Health Internal Medicine /ID# 216366, Asheboro, North Carolina
  - OnSite Clinical Solutions, LLC /ID# 216279, Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC /ID# 216368, Charlotte, North Carolina
  - Triad Clinical Trials /ID# 216792, Greensboro, North Carolina
  - Lucas Research /ID# 216487, Morehead City, North Carolina
  - Diabetes and Endocrinology Associates of Stark County Inc /ID# 216362, Canton, Ohio
  - Intend Research /ID# 216320, Norman, Oklahoma
  - Tristar Clinical Investigations PC /ID# 216944, Philadelphia, Pennsylvania
  - Frontier Clinical Research /ID# 216365, Smithfield, Pennsylvania
  - New Phase Research & Development /ID# 216774, Knoxville, Tennessee
  - Clinical Neuroscience Solutions - Memphis /ID# 216790, Memphis, Tennessee
  - Arlington Family Research Center, Inc /ID# 216363, Arlington, Texas
  - Associates in Medicine, P.A. /ID# 216781, Houston, Texas
  - FMC Science /ID# 216318, Lampasas, Texas
  - Discovery Clinical Trials-San Antonio /ID# 216866, San Antonio, Texas
  - Northwest Houston Clinical Research PLLC /ID# 216358, Tomball, Texas
  - Burke Internal Medicine & Research /ID# 216322, Burke, Virginia
  - Manassas Clinical Research Center /ID# 216313, Manassas, Virginia
  - Virginia Research Center /ID# 216341, Midlothian, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Weber MA, Aslam S, Efros MD, Chan A, Khan N, Li X, Dubcenco E, Miller MG. Single-arm study of testosterone gel replacement therapy and ambulatory blood pressure outcomes in men with hypogonadism. Andrology. 2025 Sep;13(6):1390-1401. doi: 10.1111/andr.13779. Epub 2024 Oct 9. PMID 39385523
- See also: Related Info. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants
Groups:
- AndroGel 1.62%: AndroGel 1.62% was applied topically once daily in the morning beginning at the Day 1 Visit after confirmed valid ambulatory blood pressure monitoring (ABPM) assessment and was applied at approximately the same time each day after that during the study for approximately 16 weeks. The starting dose of AndroGel 1.62% was 40.5 mg of T (2 pump actuations, applied to the upper arms and shoulders) and was titrated up or down by 20.25 mg or remained the same as assessed by morning serum T levels at Weeks 2 and 4.
Period: Overall Study
Arm/Group | AndroGel 1.62%
Started | 246
Completed | 204
Not Completed | 42
Not completed — Adverse Event | 7
Not completed — Withdrew consent | 5
Not completed — Lost to Follow-up | 9
Not completed — COVID-19 infection | 1
Not completed — Other, not specified | 20

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of study drug
Arm/Group | AndroGel 1.62%
Number analyzed (Participants) | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 246
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 209
  Black or African American | 29
  Asian | 5
  American Indian or Alaska Native | 2
  Native Hawaiian or Other Pacific Islander | 0
  Multiple | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (EOT) in 24-hour Average Systolic Blood Pressure (SBP)
Description: Systolic blood pressure was measured by the ambulatory blood pressure monitoring (ABPM) procedure. Measurements were obtained from participants using a portable data-monitoring device. The ABPM procedure was performed over a 24-hour period across 2 days and included ABPM device application by site (1st Day) and ABPM device removal by site (2nd Day).
Time Frame: Baseline, Week 16
Population: Per protocol set analysis: all participants who received at least 1 dose of study drug, were at least 85% compliant to study drug, and had valid Baseline and end of treatment systolic ABPM data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AndroGel 1.62%
Number analyzed (Participants) | 169
mmHg | 1.9 (8.99)
Statistical Analysis 1: Comparison: AndroGel 1.62%; The primary endpoint of change from Baseline to End of Treatment (EOT) in average 24-hour SBP was evaluated using a linear regression model with change in average 24-hour SBP from Baseline to EOT as the dependent variable, centralized baseline average 24-hour SBP, ongoing medical history of hypertension, and pooled study center as covariates in the per protocol population; Test type: Non-Inferiority — The hypothesis for the primary safety analysis is: H0: Change in 24-hour average SBP from Baseline to EOT ≥ 3 mmHg Vs. H1: Change in 24-hour average SBP from Baseline to EOT < 3 mmHg; LS Mean Change from Baseline to EOT = 1.9, 95% CI 2-sided [0.63 to 3.13], Standard Error of Mean 0.63

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to 30 days after the last dose of study drug; the median time on follow-up was 176 days. TEAEs and SAEs were collected from the first dose of study drug until 30 days after the last dose of study drug; mean duration on study drug was 114 days.
Arm/Group | AndroGel 1.62%
All-Cause Mortality (participants affected / at risk) | 0/246
Serious Adverse Events (participants affected / at risk) | 8/246
Other Adverse Events (participants affected / at risk) | 43/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AndroGel 1.62% (N=246)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AndroGel 1.62% (N=246)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
DIVERTICULUM GASTRIC (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
PYREXIA (General disorders) | 2 (2)
ABSCESS LIMB (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1)
INFLUENZA (Infections and infestations) | 2 (2)
OTITIS EXTERNA CANDIDA (Infections and infestations) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
LIP INJURY (Injury, poisoning and procedural complications) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 4 (4)
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 1 (1)
HEART RATE INCREASED (Investigations) | 1 (1)
LIVER FUNCTION TEST INCREASED (Investigations) | 1 (1)
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 2 (2)
GOUT (Metabolism and nutrition disorders) | 1 (1)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 2 (2)
PARAESTHESIA (Nervous system disorders) | 1 (1)
PAROSMIA (Nervous system disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
IRRITABILITY (Psychiatric disorders) | 1 (1)
DYSURIA (Renal and urinary disorders) | 1 (1)
NIPPLE PAIN (Reproductive system and breast disorders) | 1 (1)
PRIAPISM (Reproductive system and breast disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT04274894/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT04274894/SAP_001.pdf